CLINICAL TRIAL: NCT03630393
Title: Randomized Study of Ultralow Versus Standard Pneumoperitoneum Pressure During Robotic Prostatectomy Using the AirSeal® Insufflation System
Brief Title: Ultralow Versus Standard Pneumoperitoneum Pressure
Acronym: Ultralow
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: OhioHealth (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1306218
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy; Robotic; Urology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pressure 6 mmHg (Experimental): Pneumoperitoneum Pressure 6 mmHg
  Interventions: Other: Pneumoperitoneum Pressure 6 mmHg
- Pressure 15 mmHg (Active Comparator): Pneumoperitoneum Pressure 15 mmHg
  Interventions: Other: Pneumoperitoneum Pressure 15 mmHg

INTERVENTIONS:
Other: Pneumoperitoneum Pressure 6 mmHg — A pneumoperitoneum insufflation pressure of 6 mmHg will be used during robotic assisted laparoscopic prostatectomy (RALP).
  Arms: Pressure 6 mmHg
Other: Pneumoperitoneum Pressure 15 mmHg — A pneumoperitoneum insufflation pressure of 15 mmHg will be used during robotic assisted laparoscopic prostatectomy (RALP).
  Arms: Pressure 15 mmHg

SUMMARY:
The investigators plan to compare insufflation pressures during robotic assisted laparoscopic prostatectomy (RALP). Standard pressure is typically 15 mmHg, while in a previous study the investigators determined that 6 mmHg is possible routinely. Therefore, the investigators plan to compare the clinical outcomes of participants at a pneumoperitoneal pressure of 15 versus 6 mmHg.

DETAILED DESCRIPTION:
The investigators to examine the impact of low pressure during robotic assisted laparoscopic prostatectomy (RALP) with the intention of identifying whether lower pressures might benefit participants. The investigators hypothesize that a low insufflation pressure may provide an improvement in postoperative pain and abdominal distension in addition to potential physiologic benefits, and that these factors might then allow a shorter hospital stay. The investigators previously initiated a protocol in September of 2016 (IRB# 1066864) to perform RALPs at an insufflation pressure of 6 mmHg with the intention of increasing the pressure as needed on an individual participant level. In order to determine whether this might allow earlier discharge when successful, the investigators began allowing for same-day discharge in participants meeting appropriate criteria. Having now demonstrated feasibility in over 300 consecutive participants using this ultralow pneumoperitoneum protocol, the investigators now plan to conduct a randomized trial to compare a pressure of 6 mmHg with participants having RALP at a standard pressure of 15 mmHg to determine whether there is a true benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Diagnosed with prostate cancer
3. Electing to undergo robotic assisted laparoscopic prostatectomy (RALP)

Exclusion Criteria:

1. Age < 18
2. Emergency surgery
3. Patients with a significant preoperative dependence on narcotic medications
4. Unable to give informed consent
5. Dementia, history of dementia, or other significant mental impairment that would, in the opinion of the investigator, impede patient self-reporting
6. Persons participating in any other research study involving an investigational drug or device or investigational surgical procedure that could interfere with the physiologic parameters being collected (for example, a study evaluating different anesthesia regimens that could confound study results)
7. Non-English-speaking or reading

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with prostate cancer who are eligible and electing to undergo robotic assisted laparoscopic prostatectomy (RALP)
Enrollment: 170 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronney Abaza, MD, Principal Investigator — OhioHealth
Locations (1):
- Dublin Methodist Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 170 participants were consented/enrolled 31 participants were withdrawn prior to randomization (10 due to coronavirus-19 concerns; 9 due to principal investigator leaving the institution; 5 due to patient request; 3 due to change in eligibility; 3 due to resource availability; 1 at principal investigator request)
Groups:
- Pressure 6 mmHg: Pneumoperitoneum Pressure 6 mmHg
  Pneumoperitoneum Pressure 6 mmHg: A pneumoperitoneum insufflation pressure of 6 mmHg will be used during Robotic-assisted laparoscopic prostatectomy.
- Pressure 15 mmHg: Pneumoperitoneum Pressure 15 mmHg
  Pneumoperitoneum Pressure 15 mmHg: A pneumoperitoneum insufflation pressure of 15 mmHg will be used during Robotic-assisted laparoscopic prostatectomy.
Period: Overall Study
Arm/Group | Pressure 6 mmHg | Pressure 15 mmHg
Started | 68 | 71
Completed | 67 | 71
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pressure 6 mmHg: Pneumoperitoneum Pressure 6 mmHg
  Pneumoperitoneum Pressure 6 mmHg: A pneumoperitoneum insufflation pressure of 6 mmHg will be used during RALP.
- Pressure 15 mmHg: Pneumoperitoneum Pressure 15 mmHg
  Pneumoperitoneum Pressure 15 mmHg: A pneumoperitoneum insufflation pressure of 15 mmHg will be used during RALP.
- Total: Total of all reporting groups
Arm/Group | Pressure 6 mmHg | Pressure 15 mmHg | Total
Number analyzed (Participants) | 68 | 71 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (6.52) | 62.8 (6.67) | 63.5 (6.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 68 | 71 | 139
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Medication Use
Description: The cumulative dose (milligrams) of each opioid medication administered was calculated and converted to milligram morphine equivalents (MME) for each participant.
Time Frame: Through 1 week postoperatively
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Pressure 6 mmHg | Pressure 15 mmHg
Number analyzed (Participants) | 67 | 71
morphine milligram equivalents | 56.6 (40.72) | 61.2 (37.33)

2. Secondary Outcome: Post Operative Pain Scores
Description: Each participant was asked to rate their pain on a 0-10 scale, with higher numbers representing worse pain. Patients rated their pain at the following time points: in the post-anesthesia care unit (PACU) upon waking from anesthesia, at hours 4, 12, 16, and 20 after transfer to the floor, and immediately prior to discharge. The pain scores for each patient were averaged.
Time Frame: Through discharge (post-operative day 0 or post-operative day 1)
Population: Post-operative pain scores were not recorded for one participant in the Pneumoperitoneum pressure 6 mmHg group
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pressure 6 mmHg | Pressure 15 mmHg
Number analyzed (Participants) | 67 | 71
Units on a scale | 1.4 (1.61) | 1.8 (1.86)

3. Secondary Outcome: Operative Ventilation
Description: Average tidal volume (ml)
Time Frame: Intraoperatively
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Pressure 6 mmHg | Pressure 15 mmHg
Number analyzed (Participants) | 68 | 71
milliliters | 629.1 (81.9) | 629.4 (83.1)

4. Secondary Outcome: Discharge Day (Post-operative Day 0 or 1)
Description: The day of discharge (post-operative day 0 or post-operative day 1) was recorded for each participant
Time Frame: Through discharge (post-operative day 0 or 1)
Population: The post-operative discharge day was not recorded for one participant in each group
Measure: Count of Participants; unit: Participants
Arm/Group | Pressure 6 mmHg | Pressure 15 mmHg
Number analyzed (Participants) | 67 | 70
Participants
  Discharged on Post-operative day 0 | 56 | 62
  Discharged on Post-operative day 1 | 11 | 8

ADVERSE EVENTS:
Time Frame: Events were tracked through 90 days following discharge via review of medical records
Arm/Group | Pressure 6 mmHg | Pressure 15 mmHg
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/71
Serious Adverse Events (participants affected / at risk) | 1/68 | 0/71
Other Adverse Events (participants affected / at risk) | 0/68 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pressure 6 mmHg (N=68) | Pressure 15 mmHg (N=71)
Epigastric bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03630393/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03630393/ICF_001.pdf